CLINICAL TRIAL: NCT06838377
Title: Accuracy of Computer Guided Screw Holes Locating Guide and Patient Specific Champy Plate vs Conventional Champy Plate Osteosynthesis in Management of Mandibular Angle Fracture: Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed abd ellati tag eldin ahmed, general practioner dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0032025
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Mandible Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: Digital planning and custom made Champy plate manufacturing:
  Dental arches will be segmented and waxed to the ideal occlusal relationship either by mounting on semi adjustable articular or digitally. Superimposed on the CT scan using specialized software, (3Matic software Mimics-Materialize, Belgium) which also segment and realign the fracture segments virtually.
  Biomedical engineers will design the custom made Champy plate adapted on the ventral surface of the exterior oblique ridge (Champy's line of osteosynthesis) ensuring there is adequate clearance of the screw hole positions and screw lengths on the plate to avoid critical nerves, blood vessels, and adjacent teeth.
  Biomedical engineers will also design a screw hole locating device 3D printed of resin.
  The custom made Champy plate will be 3D printed in titanium using laser sintering of titanium powder (Cerea and Dolcini, 2018) with heat treatment post-processing.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided screw holes locating guide and Patient Specific Champy plate osteosynthesis (Experimental): the operation will under general anesthesia with nasal intubation and oral pack, Injection of 20 cc saline adrenaline 1:00000 to 0 in the sulcus for hemostasis, Vestibular mucosal incision, Reflect the flap to visualize the broken segments.
  Full thickness mucoperiosteal flaps were then carefully raised to expose enough underlying alveolar bone to accommodate the screw holes locating guide and the custom-made Champy plate.
  In Group I, Put the specific screw holes locating device in place and drill the screw holes, remove the screw holes locating device and mobilize the segments then apply the custom-made Champy plate and fix it with screw for passive reduction of the segments. Then suture the mucosa.
  Interventions: Device: computer guided screw holes locating guide and Patient Specific Champy plate
- conventional Champy plate osteosynthesis in management of mandibular angle fracture (Active Comparator): the operation will under general anesthesia with nasal intubation and oral pack, Injection of 20 cc saline adrenaline 1:00000 to 0 in the sulcus for hemostasis, Vestibular mucosal incision, Reflect the flap to visualize the broken segments.
  Full thickness mucoperiosteal flaps were then carefully raised to expose enough underlying alveolar bone then mobilize the broken segment, Arch bar was made to achieve proper occlusion put the Champy 2.0 plate on the ventral surface of the external oblique of the mandible and remove it for further bending using plate pliers for further accommodation of the plate then fix it in place using mono cortical screws.
  Interventions: Device: standard Champy mini plate

INTERVENTIONS:
Device: standard Champy mini plate — the operation will under general anesthesia with nasal intubation and oral pack, Injection of 20 cc saline adrenaline 1:00000 to 0 in the sulcus for hemostasis, Vestibular mucosal incision, Reflect the flap to visualize the broken segments. Full thickness mucoperiosteal flaps were then carefully raised to expose enough underlying alveolar bone then mobilize the broken segment , Arch bar was made to achieve proper occlusion put the Champy 2.0 plate on the ventral surface of the external oblique of the mandible and remove it for further bending using plate pliers for further accommodation of the plate then fix it in place using mono cortical screws.
  Arms: conventional Champy plate osteosynthesis in management of mandibular angle fracture
Device: computer guided screw holes locating guide and Patient Specific Champy plate — the operation will under general anesthesia with nasal intubation and oral pack, Injection of 20 cc saline adrenaline 1:00000 to 0 in the sulcus for hemostasis, Vestibular mucosal incision, Reflect the flap to visualize the broken segments.
  Full thickness mucoperiosteal flaps were then carefully raised to expose enough underlying alveolar bone to accommodate the screw holes locating guide and the custom-made Champy plate.
  , Put the specific screw holes locating device in place and drill the screw holes, remove the screw holes locating device and mobilize the segments then apply the custom-made Champy plate and fix it with screw for passive reduction of the segments. Then suture the mucosa.
  Arms: computer guided screw holes locating guide and Patient Specific Champy plate osteosynthesis

SUMMARY:
the aim of our study is to assess computer guided mandibular fracture reduction and to prove its lower rate of complications and higher accuracy of reduction compared to the conventional approach in management of mandibular angle fracture.

DETAILED DESCRIPTION:
This study will be conducted on 10 patients For each group selected from the Outpatient Clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Cairo University. Patients included in the study will have mandibular angle fracture indicated for open reduction and internal fixation. Patients with any systemic disease that could affect bone healing will be excluded from the study.

After accepting to be enrolled in this study, all patients will be subjected to:

I. Preoperative Assessment:

A thorough preoperative assessment of all patients will be carried out, including:

1. Dental and Medical history:

* Age
* Gender
* Health status 2. Clinical examination:
* Check vital signs (blood pressure, pulse, temperature, breathing).
* Examining soft tissue lacerations, paresthesia, swelling, hematoma. 3. Imaging:
* All patients will have DICOM CT scans with a slice thickness of 0.3-0.5 mm and covering a comprehensive field of view, encompassing the whole facial bones till the hyoid bone.
* Either silicon impressions or digital 3d scan via intraoral scanner to upper and lower dental arches are achieved.
* These scans will be used to:

  1. Diagnosis purposes: assessment of fracture: location, displaced or non-displaced, favorable or non-favorable, simple or compound or communited.
  2. Digitally segment and realign the fracture segments.

II. Digital planning and custom made Champy plate manufacturing:

Dental arches will be segmented and waxed to the ideal occlusal relationship either by mounting on semi adjustable articular or digitally. Superimposed on the CT scan using specialized software, (3Matic software Mimics-Materialize, Belgium) which also segment and realign the fracture segments virtually.

Biomedical engineers will design the custom made Champy plate adapted on the ventral surface of the exterior oblique ridge (Champy's line of osteosynthesis) ensuring there is adequate clearance of the screw hole positions and screw lengths on the plate to avoid critical nerves, blood vessels, and adjacent teeth.

Biomedical engineers will also design a screw hole locating device 3D printed of resin.

The provisional plate design will then be forwarded to the Oral and Maxillofacial Surgeon for their final approval before the digital files of the plate is sent for manufacturing.

The custom made Champy plate will be 3D printed in titanium using laser sintering of titanium powder (Cerea and Dolcini, 2018) with heat treatment post-processing.

III. Surgical procedures the operation will under general anesthesia with nasal intubation and oral pack, Injection of 20 cc saline adrenaline 1:00000 to 0 in the sulcus for hemostasis, Vestibular mucosal incision, Reflect the flap to visualize the broken segments.

Full thickness mucoperiosteal flaps were then carefully raised to expose enough underlying alveolar bone to accommodate the screw holes locating guide and the custom-made Champy plate.

In Group I, Put the specific screw holes locating device in place and drill the screw holes, remove the screw holes locating device and mobilize the segments then apply the custom-made Champy plate and fix it with screw for passive reduction of the segments. Then suture the mucosa.

In Group II, mobilize the broken segment first, Arch bar was made to achieve proper occlusion put the Champy 2.0 plate on the ventral surface of the external oblique of the mandible and remove it for further bending using plate pliers for further accommodation of the plate then fix it in place using mono cortical screws.

IV. Evaluation protocol Scheduled follow-up intervals were 1, 2, 4, 8 and 12 weeks postoperatively. Postoperative complications, defined as a need for further intervention, were detailed prospectively over a period of at least 6 months postoperative.

Radiographic assessment will be achieved by CT scan preoperatively and postoperatively within one week to assess the following:

* to calculate any amount for segments deviation from the virtual plan in mms.
* For prevention of complications: hematoma, swelling, dehiscence and infection.

V. Statistical Methods:

* Descriptive statistics, including means and standard deviations, will be calculated to summarize the data. The statistical analysis will be performed using SPSS statistical software version 22 (IBM, Armonk, NY). The analysis will be conducted by a single statistician from Cairo University, cairo, Egypt.
* For the evaluation of primary and secondary outcomes, the chi-square statistic will be used. A significance level (p-value) of less than 0.05 will be considered statistically significant, indicating a significant difference between groups or variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated mandibular angle fracture needs open reduction and internal fixation.
* Patients with medical history that did not hinder plate placement and adequate proper oral hygiene.
* Both genders males and females will be included.

Exclusion Criteria:

* General contraindications to surgery. .
* Patients with comminuted fractures.
* Subjected to irradiation in the head and neck area less than 1 year before fixation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Patients participating in other studies, if the present protocol could not be properly followed.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of computer guided screw holes locating guide and Patient Specific Champy plate in management of mandibular angle fracture | 3 months
  calculate any amount for segments deviation from the virtual plan in mms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt